CLINICAL TRIAL: NCT03483818
Title: A Pilot Trial of Directly Observed Anti HCV Therapy Supported With Contingency Management in a Population on Opiate Substitute Therapy
Brief Title: Pilot Trial of Directly Observed Anti HCV Therapy & Contingency Management in a Population on Opiate Substitute Therapy
Acronym: DOT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Collaborators: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014CO01
Record Dates: First submitted 2015-11-27; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2017-12

CONDITIONS: Hepatitis C
Keywords: Community Pharmacy; Antiviral Therapy
MeSH Terms: conditions — Hepatitis C | interventions — Restraint, Physical; Antiviral Agents

STUDY DESIGN:
Intervention Model Description: This is a feasibility study comparing delivery of care pathways rather than evaluating medication
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist-Led Pathway (Active Comparator): Assessment & Treatment of HCV infection with oral antivirals in a community pharmacy pathway
  Interventions: Procedure: Assessment & Treatment of HCV infection with oral antivirals
- Conventional Care Pathway (Active Comparator): Assessment & Treatment of HCV infection with oral antivirals in a conventional care pathway
  Interventions: Procedure: Assessment & Treatment of HCV infection with oral antivirals

INTERVENTIONS:
Procedure: Assessment & Treatment of HCV infection with oral antivirals — This is a cluster randomised trial of directly observed anti HCV therapy versus conventional care in HCV positive patients, who are in a pharmacist delivered OST program, where the patients attending an individual pharmacist are the cluster. Pharmacies participating in the trial will be allocated to conventional care pathway or the pharmacist-led pathway.

SUMMARY:
DOT-C is a cluster randomised trial of a pharmacist-led, directly observed anti HCV therapy pathway versus the conventional care pathway within community pharmacies. The primary trial outcome is to evaluate the effect of pharmacist-led anti-HCV directly observed therapy on the proportion of patients reaching a sustained virological response.

DETAILED DESCRIPTION:
DOT-C is a cluster randomised trial of a pharmacist-led, directly observed anti HCV therapy pathway versus the conventional care pathway within 8 community pharmacies. Patients attending an individual pharmacy are the cluster. Pharmacies who are participating in the trial will be allocated to the pharmacist-led pathway or the conventional care pathway. The pilot trial aims to recruit 40 patients into the both the pharmacist-led and the conventional care pathways.

Approximately 2,000 patients are prescribed OST within the Tayside region of North East Scotland. Around 85% of these patients receive daily or regular supervision of their OST consumption through one of the 92 community pharmacies. It is expected that at least 40% of these patients will be infected with HCV and that around 40% of infections will be with Genotype 1 virus. The 8 pharmacies acting as cluster sites for this trial have around 400 patients attending for supervised OST administration.

Design: This is a cluster randomised trial of directly observed anti HCV therapy versus conventional care in HCV positive patients, who are in a pharmacist delivered OST program, where the patients attending an individual pharmacist are the cluster. Pharmacies participating in the trial will be allocated to conventional care pathway or the DOT pathway.

Entry into the trial will be following a positive HCV test at which stage the patient will be allocated to a pathway, dependent on the pharmacy they are attending. The pathways are:

* Pharmacy DOT
* Conventional care pathway

Research Questions Trial

1. Does a pharmacist-led HCV treatment pathway increase the uptake of testing and treatment by OST users and result in a higher proportion of patients achieving a sustained virological response (SVR) compared to the conventional pathway?
2. Can a pharmacist-led pathway be introduced in a way that is feasible and acceptable to users and service providers and are there any unintended consequences?

Conventional Care Pathway In pharmacies randomised to the conventional care pathway, the pharmacist will opportunistically discuss with the patient the possibility of HCV infection. Information will be provided verbally and by offering standard leaflets about HCV and local services for testing and or treatment. Patients who seek referral for testing and/or treatment will be managed according to the standard local treatment pathway. The pharmacist will record on a screening log which OST patients they have had the discussion with. If the patient achieves a referral and attends treatment at one of the dedicated treatment centres, the treatment nurses will enquire about any methadone prescription and which pharmacy is providing the methadone. The participant's medical regimen will be as standard but that there will be some additional data collection. As this is a real world study patients may be referred into treatment by other agencies (e.g. drug keyworker) after a positive test; if tested within pharmacy their data will be captured for this study.

Pharmacist-Led Pathway In pharmacies randomised to the Pharmacist pathway, the staff training and educational materials on HCV testing, HCV treatment, and behaviour change will be delivered. At the start of the pathway pharmacists will discuss HCV infection with their OST patients. Those with unknown HCV status will be offered testing using DBS in the pharmacy. In pharmacies where dried blood spot testing for HCV is not available this will be established. Patients identified as HCV positive will have a post-test discussion with the pharmacist. During this discussion the pharmacists will obtain informed consent, explain about HCV treatment. Next, the pharmacist will offer them anti-HCV therapy in the pharmacy. The patients who decline study participation will be entered in the screening log. For the patients who do consent, the pharmacist will complete a pre-treatment checklist of medical co-morbidities, medical history, concomitant medication to look for drug-drug interactions, and blood tests including viral parameters. This will also include a set of blood tests to check full blood count, urea and electrolytes, liver function testing, including markers of liver fibrosis (Fib4, APRI, AST:ALT ratio) and viral parameters (genotype and load), this will be performed outside the pharmacy at a local health care facility that provides a routine phlebotomy service. These bloods are standard of care for HCV treatment and are not research specific (i.e., they are also part of the Conventional pathway). If there are no contra-indications to therapy, the patient will commence the treatment. In patients where there are contraindications or queries about suitability, the pharmacist will contact the central clinical co-ordinator for advice. Unsuitable patients will be referred to local hospital services for assessment outside the study as standard clinical care. The suitable patients entering treatment will have daily dispensing of therapy drugs with consumption of antivirals observed at the same time as the OST within the pharmacy (usually 5 or 6 days, so a modified version of DOT). For doses that patients have to self-administer and the weekend doses when there is no OST distribution), the pharmacist and patient will make a brief if-then action plan (an implementation intention) and coping plan (to overcome anticipated barriers)(19).

Recruitment Patients in OST attending participating pharmacies will be recruited after a new HCV diagnosis or patients with a previous known diagnosis would be systematically approached to participate in the trial. Those that agree to enter the trial would provide consent and at this point be randomised to the different pathways dependent on the pharmacy they are attending. For the study there would be no further adjustment of the groups so the trial will be testing the whole pathway of care.

For those patients attending a pharmacy within the DOT cluster, a Pharmacist-led, protocol-driven checklist for therapy suitability, with medical review available for participants who fall outside protocol, would be performed.

Consenting Participants Potential participants will be approached by pharmacy staff familiar with the trial methodology and trained in obtaining informed consent in clinical trials.

Randomisation Eight pharmacies will be enrolled to this study. They will be split into two matched groups based on geography and patient numbers. Four will be allocated to pharmacist DOT. The four pharmacies allocated to conventional care will refer patients to the local BBV services. Randomisation will be carried out using http://www.randomization.com . The subjects are randomized into 1 block. To reproduce this plan, use the seed 12576 along with the number of subjects per block/number of blocks and (case-sensitive) treatment labels as entered above.

Intervention Allocation All participants will have HCV testing and genotyping and will be allocated to conventional BBV treatment based on the HCV genotype. Only those patients who are genotype 1 will be enrolled in this study. Participants will be allocated to pharmacist led or conventional pathway; contingency management or not, according to the cluster pharmacy that they normally use.

Sample Size - Since this a pilot study no sample size calculation has been performed Overview of Qualitative Research Components The qualitative research will take the form of a process evaluation designed to inform aspects of the proposed phase III trial. It will contribute to assessing the feasibility and acceptability to service users and service providers of using pharmacies to deliver testing and treatment alongside OST delivery (including identification of barriers and facilitators); identifying any unintended consequences of participation; exploring responses to randomization approaches; providing guidance on how the intervention might be modified for the Phase III randomised controlled trial.

Interviews will be conducted with small samples of (i) service users and (ii) relevant professionals. This work will expand on qualitative research already undertaken with clients and professionals in the pilot work and modelling that preceded this study. Qualitative interviews will be conducted with service users and professionals using semi-structured topic guides developed in line with the research aims. Topics will not be explored in a prescriptive manner but as part of an open discussion. This flexible format will enable additional salient topics and insights to emerge. In broad terms, the focus for the different respondent groups will be as follows:

Health Economic Assessments - Economic analysis will be undertaken alongside the trial, utilising the costs, resource use and effectiveness data generated within the trial. For example, the cost service delivery, staff time, will be collected and combined with other resource use data. The number of patients achieving SVR at the end of the trial will be combined with the cost data to calculate the incremental cost per cure for each pathway.

This phase II trial will establish a workable design and approach in order to reduce the risks associated with a future definitive phase III multicenter randomized controlled trial and establish a framework to assess the costs and benefits of using a community pharmacy pathway to treat HCV in patients participating in an OST program

ELIGIBILITY:
Inclusion Criteria:

* HCV PCR positive to genotype 1
* On Opioid Substitution Therapy dispensed and with supervised administration by pharmacist

Exclusion Criteria:

* HCV PCR positive to any genotype other than genotype 1
* Evidence of current or previous decompensated liver disease
* HIV infection
* HBsAg positive with detectable HBV DNA
* Aggressive or violent behaviour
* Inability to provide informed consent
* Pregnancy or breast feeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The number of patients reaching a sustained virological response in the pharmacist -led arm, as compared with the current treatment pathway for patients receiving opiate substitution therapy | Sustained Virological response will be assessed at 12 weeks post completion of therapy
  Participants who complete the pathway and undertake a test for viral clearance

SECONDARY OUTCOMES:
Cost effectiveness of the pharmacist DOT pathway as compared with the conventional care pathway | One Year post trial completion
  The cost profile of elements of pathway delivery
Comparison of rate of HCV testing rates in pharmacist pathway compared with current pathway | Sustained Virological response will be assessed at 12 weeks post completion of therapy
  The number of participants agreeing to take a dried blood spot test compared to the available pool of patients

CONTACTS AND LOCATIONS:
Overall Officials: John Dillon, Study Director — NHS Tayside
Locations (1):
- Ninewells Hospital, Dundee, Tayside, United Kingdom

REFERENCES:
- [Result] Radley A, Tait J, Dillon JF. DOT-C: A cluster randomised feasibility trial evaluating directly observed anti-HCV therapy in a population receiving opioid substitute therapy from community pharmacy. Int J Drug Policy. 2017 Sep;47:126-136. doi: 10.1016/j.drugpo.2017.05.042. Epub 2017 Jun 21. PMID 28647161
- See also: Publication of study outcomes — https://doi.org/10.1016/j.drugpo.2017.05.042